CLINICAL TRIAL: NCT06225219
Title: Establishing the Chaplain Role in a Primary Care Clinic Setting
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 024.CHP.2022.D
Record Dates: First submitted 2023-11-13; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Emotional Disorder
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Counseling — To introduce a model of holistic care to the patient populations served by the GCAC through chaplain interventions that focus on spiritual and emotional health.
  Other Names: Chaplain interventions; Model of holistic care

SUMMARY:
In 2019, a full-time chaplain was placed in the Golden Cross Academic Clinic (GCAC), with the chaplain's focus being in the primary care internal medicine department. While research exists regarding chaplains in the inpatient setting, research regarding the presence of a full-time chaplain in a primary care setting as well as the topics patients discuss with that chaplain are limited.

DETAILED DESCRIPTION:
A few studies conducted in the hospital setting have shown what topics patients typically discuss with a chaplain. In the article, "Patients and Loved Ones' Expectations of Chaplain Services. Munchausen and colleagues present that the two highest-rated services performed by chaplains were spiritual and emotional support. This study also found that patients wanted to see a chaplain for the following reasons: to be listened to, to be with in times of anxiety, to offer support to loves ones, to remind of God's care and presence, to pray, for religious rituals, to assist with the understanding of advance care planning documents, and to counsel regarding moral or ethical decisions.

ELIGIBILITY:
Inclusion Criteria:

* • Patient at the GCAC who are > 18 years old

  * Met with a member of the on-staff chaplaincy during a visit to GCAC

Exclusion Criteria:

* • Patient did not meet with a member of the on-staff chaplaincy during a visit to GCAC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient at the GCAC who are > 18 years old
  • Met with a member of the on-staff chaplaincy during a visit to GCAC
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
Number of times chaplain is requested by patient or provider | 1 year
  Number of request from the patients or provider for chaplain
Usefulness, feasibility, and reception of screening mechanism for GCAC staff | 1 year
  Develop a screening mechanism that allow GCAC staff to identify patients who could benefit from spiritual and emotional support.
Themes discussed during meeting between chaplain and patient | 1 year
  Explore themes from patient conversations with a chaplain
Number of meetings/conversations pertaining to each theme identified | 1 year
  Theme identified for the number of meetings/conservations

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dowden, PhD, Principal Investigator — Methodist Midlothian Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years